CLINICAL TRIAL: NCT04424498
Title: Absorbable Rods and Kirschner Wires for the Treatment of Displaced Radial Neck Combined With Olecranon Fractures in Children
Brief Title: Treatment of Displaced Radial Neck Combined With Olecranon Fractures
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuxi Su, Vice professor, Children's Hospital of Chongqing Medical University
Other Study IDs: CQMU20200016
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Child
Keywords: Kirschner wires; Absorbable rods; Radial neck fracture; Olecranon fracture
MeSH Terms: conditions — Radial Head and Neck Fractures; Olecranon Fracture | interventions — Bone Wires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Absorbable Rods and Kirschner Wires — A Boyd incision was applied in all patients; olecranon fractures were reduced first and fixed with Kirschner wires. Then, the displaced radial neck fractures were reduced and fixed using absorbable rods.

SUMMARY:
This study aimed to evaluate the outcomes of using absorbable rods and Kirschner Wires technique for severe displaced radial neck fractures combined with olecranon fractures in children.

DETAILED DESCRIPTION:
The most common fracture in children is the elbow fracture, and the three most common elbow fractures are supracondylar, lateral condylar, and medial epicondylar fractures. Elbow fractures are easy to diagnose and the treatment modalities are studied often. However, proximal radius fractures, which include radial neck and head fractures, remain challenging to diagnose and manage. In addition, proximal radius fractures are often combined with other fractures, most commonly, an olecranon fracture. Most radial neck fractures can be treated conservatively if the displacement is less than 3 mm and the angle is less than 30º. However, for severe Judet type III and type IV radial neck fractures, surgery is inevitable.

This study focused on radial neck fractures combined with an olecranon fracture. In this study, absorbable rods were used for fixation of radial head fractures, and with no need for removal of the inner fixation, we performed anatomy reduction via the same incision with direct vision of the olecranon, and we were able to fix the fractures with Kirschner wires (K-wires). In this retrospective study, we aimed to evaluate a treatment method for severe displaced radial neck combined with olecranon fractures in children using a Boyd incision, absorbable rods, and K-wires.

ELIGIBILITY:
Inclusion Criteria:

* open reduction of severe radial neck fractures combined with an olecranon fractures in the same elbow
* fixation performed using absorbable rods and K-wires

Exclusion Criteria:

* single radial head fractures or single olecranon fractures
* fixation performed with bands
* old fractures,
* Boyd incision was not used,
* guardians did not agree with the surgery

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Medical records of patients who attended our hospital between Jan 2012 and Dec 2016 were retrospectively reviewed.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Mayo Elbow Performance Index score | 3th month after surgery
  MEPI results were categorized as follows: >90 points, excellent; 81-90 points, good; 61-80 points, fair; and <60 points, poor.

CONTACTS AND LOCATIONS:
Overall Officials: Yuxi Su, M.D., Principal Investigator — Children's hospital of Chongqing Medical Univeristy
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No